CLINICAL TRIAL: NCT01467362
Title: Efficacy of the V0034CR01B Emollient on Xerosis in Children With Atopic Dermatitis. Randomised, Vehicle-controlled, Parallel-groups, Double-blind Study With an Open Label Extension.
Brief Title: Efficacy Emollient on Xerosis in Children With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V00034 CR 3 12 1B; 2011-003295-37 (EudraCT Number)
Record Dates: First submitted 2011-10-24; First posted 2011-11-08 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Atopic Dermatitis
Keywords: xerosis; dry skin; dermatitis; pruritus; eczema; emollient; corticosteroid
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Pruritus; Eczema | interventions — Desonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- V0034CR01B (Experimental)
  Interventions: Drug: V0034CR01B; Drug: desonide 0.1% cream; Other: Foaming gel
- Vehicle cream (Placebo Comparator)
  Interventions: Drug: Vehicle cream; Drug: desonide 0.1% cream; Other: Foaming gel

INTERVENTIONS:
Drug: V0034CR01B — Cream Out of flares: 1 application bid (morning and evening) During flares: 1 application once a day (in the morning) Maximum 91 days
  Arms: V0034CR01B
Drug: Vehicle cream — Cream Out of flares: 1 application bid (morning and evening) During flares: 1 application once a day (in the morning) Maximum 28 days
  Arms: Vehicle cream
Drug: desonide 0.1% cream — cream, once a day (in the evening) during flares
  Other Names: Locapred
Other: Foaming gel — for the washing and cleaning
  Other Names: Pediatril

SUMMARY:
Atopic dermatitis is a frequent, chronic inflammatory disease influenced by local, immunological, genetic and environmental factors. Important symptoms of atopic dermatitis are dry skin, intense pruritus and impaired epidermal barrier function. Atopic dermatitis is associated with skin barrier dysfunction that facilitates an easier allergen penetration into the skin with an increased irritation and subsequent cutaneous inflammation. A lack of important stratum corneum intercellular lipids and an inadequate ratio between compounds enhance trans-epidermal water loss leading to xerosis. Skin hydration by emollient therapy usually twice daily improves dryness and subsequently pruritus during the treatment of atopic dermatitis and especially improves the barrier function. Emollients make part of basic therapy (grade 1) for treatment of atopic dermatitis (European Academy of Dermatology and Venereology Task Force 2009 Position Paper). Improvement of cutaneous barrier alteration, measured by skin hydration, is a key element for evaluation of emollient treatment efficacy.

The primary objective of this study is to demonstrate the efficacy of the tested product (V0034CR01B) cream on xerosis in children with atopic dermatitis compared to the excipient formula during 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with atopic dermatitis, dry skin, objective SCORAD < 15,
* With xerosis on the body and a xerosis score > = 2 (SCORAD sub-score) on the anterior part of lower limbs,

Exclusion Criteria:

* Acute phase of atopic dermatitis
* Severe form of atopic dermatitis

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 251 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Xerosis score: mean evolution over the different time-points of double-blind period | During 28 days (Day 1, Day 7, Day 14, Day 21 and Day 28)

SECONDARY OUTCOMES:
Hydration Index score : measurement of the skin hydration | Day 1, Day 14, Day 28, Day 56 and Day 84
Xerosis score evolution over the different time-ponts during open label period | At Visit1 (Day 1) and at Day 56 and Day 84
Xerosis Visual Analogue Scale (evaluation skin dryness) | Day 1, Day 14, Day 28, Day 56 and Day 84
Scoring for Atopic Dermatitis (SCORAD) : measurement of objective symptoms of Atopic Dermatitis. | Day1, Day 28, Day 56 and Day 84.
Overall assessment of treatment efficacy by the investigator | Day 28 and Day 84
Overall assessment of treatment efficacy and use by the parent(s)/guardian(s) | at Day 28 and at Day 84
Assessment of the local tolerability and the systemic safety (reported adverse events) | Day 1, Day 7, Day 14, Day 21, Day 28, Day 56 and Day 84
Topical corticosteroid assessment | Day 7, Day 14, Day 21, Day 28, Day 56 and Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Franck BORALEVI, Pr, Principal Investigator — Health centre
Locations (25):
- Estonia (2):
  - Estonia, Tallinn
  - Estonia, Tartu
- France (5):
  - France, Bordeaux
  - France, Martigues
  - France, Nantes
  - France, Nice
  - France, Poitiers
- Lithuania, Vilnius, Lithuania
- Poland (9):
  - Poland, Bialystok
  - Poland, Inowrocław
  - Poland, Lodz
  - Poland, Oleśnica
  - Poland, Poznan
  - Poland, Płock
  - Poland, Strzelce Opolskie
  - Poland, Warsaw
  - Poland, Żyrardów
- Romania (8):
  - Romania, Brasov
  - Romania, Bucharest
  - Romania, Constanța
  - Romania, Craiova
  - Romania, Iași
  - Romania, Ploieşti
  - Romania, Sibiu
  - Romania, Târgu Mureş